CLINICAL TRIAL: NCT00445588
Title: A Phase II Trial of Erlotinib (OSI-774) and Sorafenib (BAY 43-9006) for Patients With Progression or Recurrent Glioblastoma Multiforme
Brief Title: Erlotinib and Sorafenib in Treating Patients With Progressive or Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03018; NCI-2012-03018 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR531731; NABTT 0502 (Other: New Approaches to Brain Tumor Therapy Consortium); NABTT-0502 (Other: CTEP); U01CA062475 (NIH)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Erlotinib Hydrochloride; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Patients receive oral erlotinib hydrochloride 150mg once daily and oral sorafenib tosylate 400mg twice daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study
  Interventions: Drug: erlotinib hydrochloride; Drug: sorafenib tosylate; Other: pharmacological study

INTERVENTIONS:
Drug: erlotinib hydrochloride — 150mg Given orally once daily
  Other Names: OSI-774
Drug: sorafenib tosylate — 400mg Given orally twice daily
  Other Names: BAY 3-9006
Other: pharmacological study — Correlative studies

SUMMARY:
This phase II trial is studying how well giving erlotinib together with sorafenib works in treating patients with progressive or recurrent glioblastoma multiforme. Erlotinib and sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving erlotinib together with sorafenib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this trial is to estimate the overall survival rate associated with this combined regimen in treating adult patients with recurrent glioblastoma multiforme.

SECONDARY OBJECTIVES:

I. To assess and estimate the toxicities. II. Tumor response rate. III. To estimate 6-month progression free survival. IV. To describe the pharmacokinetics of this route of administration. V. For the Molecular Targeted Combinations Correlative (MTC2) Study Initiative: To determine the relationship between tumor and blood biomarkers and clinical outcome of patients treated with the combination of targeted agents.

OUTLINE: This is a multicenter, open-label, phase II study.

Patients receive oral erlotinib hydrochloride once daily and oral sorafenib tosylate twice daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Tumor tissue and blood samples are collected prior to beginning treatment. Samples are analyzed by immunohistochemistry, gene expression, and DNA mutation and genomic analyses of the epidermal growth factor receptor, ras-raf-ERK, and PI3K-Akt-mTOR pathways to identify markers that correlate with patient outcomes. Blood samples are also collected on day 15 of course 1 for pharmacokinetic studies. Samples are analyzed by reversed-phase isocratic high-performance liquid chromatography with electrospray ionization mass spectrometry to determine the concentration of erlotinib hydrochloride and sorafenib tosylate and its known metabolites.

After completion of study therapy, patients are followed every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed supratentorial glioblastoma multiforme which is progressive or recurrent after radiation therapy ± chemotherapy; patients with previous low grade glioma who progressed after radiotherapy ± chemotherapy and are biopsied and found to have a high grade glioma are eligible
* Patients must have tissue specimens available and agree to have their blood and tissue blocks (or slides) submitted for the combined correlative studies
* Patients must have measurable contrast enhancing progressive or recurrent glioblastoma multiforme by MRI or CT imaging (Within 14 days before starting treatment)
* Patients must have recovered from toxicity of prior therapy. An interval of at least 3 months must have elapsed since the completion of the most recent course of radiation therapy, while at least 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen, and at least 6 weeks since the completion of a nitrosourea containing chemotherapy regimen; NOTE: For a non-cytotoxic, FDA approved agents (i.e. Celebrex, thalidomide, etc.) therapy could be started 2 weeks after discontinuing this agent provided the patient has fully recovered from all toxicity associated with the agent; for investigational, non-cytotoxic agents a minimum of 3 weeks must have elapsed before the patient will be eligible for this study
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute Neutrophil Count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Creatinine =< 1.7mg/dl
* Total Bilirubin within normal institutional limits
* Transaminases =< 2.5 times above the upper limits of the institutional norm
* PT, PTT ≤ institutional norm
* Patients must be able to provide written informed consent
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception; women of childbearing potential must have a negative serum pregnancy test; (the anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant)
* Patients must have a Mini Mental State Exam score >= 15

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety; (examples of medical illnesses are [but not limited to] the following: uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements)
* Patients with uncontrolled hypertension; hypertension with systolic blood pressure of > 140 mmHg or diastolic pressure > 90 mmHg; however, patients with well-controlled hypertension are eligible
* Patients who are pregnant or breast-feeding (the anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant)
* Patients who have received more than two prior treatments
* Patients who have had prior therapy with erlotinib or sorafenib or any other agent targeting EGFR
* Patients receiving concurrent therapy for their tumor (with the exception of steroids)
* Patients undergoing major surgery or sustaining a significant traumatic injury within 21 days prior to treatment are ineligible
* Patients with a concurrent malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin; patients with a prior malignancy are ineligible unless they have been free of disease for >= five years
* Patients must not have any evidence of bleeding diathesis or coagulopathy
* Patients with PT INR > 1.5 are excluded, unless the patient is on full dose warfarin
* Patients on full-dose anticoagulants (e.g., warfarin) are eligible provided that both of the following criteria are met:

  * The patient has an in-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * The patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
  * NOTE: Patients on a full dose of anticoagulants will a different schedule for PT/INR evaluations
* Prophylactic anticoagulation (i.e. low dose warfarin) are eligible provided their coagulation parameter levels are as follows: prothrombin time (INR; International Normalized Ratio of prothrombin time) < 1.1 x institutional upper limit of normal
* Patients with known abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test) are excluded
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow pills are excluded
* Patients cannot be receiving cytochrome P450-inducing anticonvulsants (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital, primidone, oxcarbazepine) and must not have taken them for at least 10 days
* Patients may not have allergies to or a history of allergic reactions attributed to erlotinib and/or sorafenib
* Eligibility of patients receiving any other medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of erlotinib or sorafenib will be determined following review of their case by the Principal Investigator
* HIV patients receiving combination anti-retroviral therapy will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — New Approaches to Brain Tumor Therapy Consortium
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Peereboom DM, Ahluwalia MS, Ye X, Supko JG, Hilderbrand SL, Phuphanich S, Nabors LB, Rosenfeld MR, Mikkelsen T, Grossman SA; New Approaches to Brain Tumor Therapy Consortium. NABTT 0502: a phase II and pharmacokinetic study of erlotinib and sorafenib for patients with progressive or recurrent glioblastoma multiforme. Neuro Oncol. 2013 Apr;15(4):490-6. doi: 10.1093/neuonc/nos322. Epub 2013 Jan 17. PMID 23328813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult pts accured in an outpatient clinic between Jan 2007 and October 2007.
  pts had to have measurable , histologically proven GBM, that had progressed following radiation therapy and 0-2 prior chemotherapies.
Groups:
- Treatment: Patients receive oral erlotinib hydrochloride 150 mg once daily and oral sorafenib tosylate 400 mg twice daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study
  erlotinib hydrochloride 150mg: Given orally once daily
  sorafenib tosylate 400mg: Given orally twice daily
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Treatment
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: histologically confirmed GBM, progressed or recurred following RT and 0-2 prior chemotherapy regimens
Groups:
- Treatment: Patients receive oral erlotinib hydrochloride 150mg once daily and oral sorafenib tosylate 400mg twice daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study
  erlotinib hydrochloride: 150mg Given orally once daily
  sorafenib tosylate: 400mg Given orally twice daily
  pharmacological study: Correlative studies
Arm/Group | Treatment
Number analyzed (Participants) | 56
Age, Continuous [Median (Full Range); unit: years] | 56 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 35
Karnosky Performance Status [Number; unit: participants] — 100 - Normal; no complaints; no evidence of disease 90 - Able to carry on normal activity; minor signs or symptoms of disease 80 - Normal activity with effort; some signs or symptoms of disease 70 - Cares for self; unable to carry on normal activity or to do active work 60 - Requires occasional assistance, but is able to care for most of his personal needs
  participants
    90-100 | 26
    60-80 | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: death. measured by time of first day of treatment until date of death, assessed up to 2 years.
Time Frame: Time of first day of the treatment to death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment: Patients receive oral erlotinib hydrochloride 150mg once daily and oral sorafenib tosylate 400mg twice daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Other: pharmacological study
  erlotinib hydrochloride 150mg: Given orally once daily
  sorafenib tosylate 400mg: Given orally twice daily
  pharmacological study: Correlative studies
Arm/Group | Treatment
Number analyzed (Participants) | 56
months | 5.7 [4.5 to 7.9]
Statistical Analysis 1: Comparison: Treatment; The overall failure rate will be estimated by dividing the number of events (death) with the total exposure time in the study cohort. 95% confidence intervals and median time of survival will be calculated using standard methods; Test type: Superiority or Other; p = 0.4, Regression, Cox — cox regression model was used to estimate the HR of death compared to NABTT historical control with same histology, adjusted for age, KPS, and surgical procedure; cox regression model used to estimate the HR of death compared to NABTT historical control same histology, adjusted for age, KPS, surgical procedure; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.6 to 1.3]

2. Secondary Outcome: 6months -Progression-free Survival Rate
Description: defined patient started treatment is alive and progression free at the time of 26-week (6 months) follow-up
Time Frame: At 6 months- defined as patient started treatment is alive and progression free at the time of 26-week (6 months) follow-up
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 56
percentage of participants | 14 [8 to 28]

ADVERSE EVENTS:
Time Frame: events collected from first day of dosing till off treatment - approximately 2 years
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 9/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=56)
fatigue (General disorders) | 5 (5)
lipase increased (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less